CLINICAL TRIAL: NCT02550613
Title: Evaluation of Treatment Response With Integrated MRI/PET in Patients With Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201401081MIND
Record Dates: First submitted 2015-09-14; First posted 2015-09-15 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: MR/PET, hepatocellular carcinoma, HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: The imaging biomarkers determined by MR-PET — The purpose of this study is to explore the ability of integrated MRI/PET to detect and evaluate treatment outcome in HCC patients. This study using 18F-FDG PET and functional MRI (DCE-MRI, Diffusion-weighted MRI, MR spectroscopy).

SUMMARY:
The purpose of this study is to explore the ability of integrated MRI/PET to detect and evaluate treatment outcome in HCC patients.

DETAILED DESCRIPTION:
This study using 18F-FDG PET and functional MRI (DCE-MRI, Diffusion-weighted MRI, MR spectroscopy).

ELIGIBILITY:
Inclusion Criteria:

1. Prior Informed Consent Form
2. At least one measurable tumor, according to RECIST version 1.1.
3. Age > 20 years.
4. ECOG performance status 0 or 1.
5. Life expectancy > 3 months.
6. Confirmed Diagnosis of HCC
7. Adequate renal function (Serum creatinine ≦ 1.5 x upper limit of normal).

Exclusion Criteria:

1. Age <20 years old
2. Pregnancy
3. Contraindication for MRI: claustrophobia or MR non-compatible devices
4. Contraindication for MR contrast medium: severe adverse reaction or impaired renal function (Cre > 2.0)
5. History of other malignancy

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll 100 HCC patients who are admitted for curative or non-curative treatments, including operation, radiofrequency ablation, TACE, target therapy, chemotherapy, or radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-05; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
The recurrence rate at 3 months after treatment | 3 months

SECONDARY OUTCOMES:
The overall survival after treatment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bang-Bin Chen, MD, Principal Investigator — Department of Medical Imaging, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan